CLINICAL TRIAL: NCT00974870
Title: A Split-face Randomized Controlled Trial to Assess the Efficacy of a Needling Device for the Treatment of Acne Scars
Brief Title: A Pilot Study Testing the Efficacy of a Needling Device for the Treatment of Acne Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology- Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU15904
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Acne Scars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- needling treatment (Experimental): Needling treatment applied to half of the face at each study visit
  Interventions: Procedure: needling treatment
- Control (No Intervention): No treatment applied to half of the face

INTERVENTIONS:
Procedure: needling treatment — Needling treatment applied to half of the face at each study visit
  Arms: needling treatment

SUMMARY:
The primary objective of this study is to determine the efficacy of a needling device for treatment of acne scars.

DETAILED DESCRIPTION:
We are investigating a needled micro-roller for use in improving the appearance of acne scars. The study is being conducted under the direction of Dr. Murad Alam of Northwestern University, Department of Dermatology.

The needles on the micro-roller are designed to create small holes in the top and mid layers of skin in order to induce the formation of more collagen, which would in turn help improve the appearance of acne scars. To qualify for the study, you must have at least 2 large areas of the face with acne scars.

The study is designed such that one part of your face, which has acne scars, will be treated with the device on 3 separate occasions, spaced 2 weeks apart at our clinic in Chicago at Northwestern. We would also ask you to return at 3 months and at 6 months to have photographs taken.

If you are interested in participating, we would like to get you involved as soon as possible

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70 years old
* Subjects in general good health
* The subject has the willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator
* Global Acne Scarring Classification grade 2-41 (Appendix II)
* Subject has at least two areas of acne scaring on the face (with at least 2 acne scars in each) that are at least 2 cm apart

Exclusion Criteria:

* Pregnancy and lactation
* Subjects with history of keloid or hypertrophic scars
* Subjects with active skin disease (other than mild acne) or skin infection in the treatment area
* Subjects with an active systematic or local skin disease that is likely to alter wound healing
* Subjects who have undergone in the past 6 months or planning to undergo in the next 6 months the following cosmetic treatments in the acne scar area

  * Injectable permanent filler
  * Ablative laser treatment
* Subjects taking the following prescription medications:

  * Accutane or other retinoids within the past 12 months
  * Anticoagulant (warfarin)
* Subjects who allergic to lidocaine and prilocaine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
We will evaluate qualitatively and quantitatively the improvement of the subject's acne scars | 6 months

SECONDARY OUTCOMES:
The tolerability of the treatment will be assessed | 4 weeks
Subject satisfaction will be determined | 6 months
Any adverse events of this treatment will be recorded. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Derived] Alam M, Han S, Pongprutthipan M, Disphanurat W, Kakar R, Nodzenski M, Pace N, Kim N, Yoo S, Veledar E, Poon E, West DP. Efficacy of a needling device for the treatment of acne scars: a randomized clinical trial. JAMA Dermatol. 2014 Aug;150(8):844-9. doi: 10.1001/jamadermatol.2013.8687. PMID 24919799